CLINICAL TRIAL: NCT00458913
Title: Phase II Study of Bortezomib (VELCADE) With Cisplatin as First Line Treatment of Malignant Mesothelioma
Brief Title: Bortezomib and Cisplatin as First-Line Therapy in Treating Patients With Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-08052; JJPRD-26866138CAN2012; 2006-000009-51 (EudraCT Number)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; recurrent malignant mesothelioma; advanced malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Bortezomib; Cisplatin

INTERVENTIONS:
Drug: bortezomib
Drug: cisplatin

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with cisplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving bortezomib together with cisplatin works as first-line therapy in treating patients with malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity and safety of bortezomib and cisplatin as first-line treatment in patients with malignant mesothelioma.
* Validate the use of progression-free survival rate as a primary endpoint for the design of phase II mesothelioma trials.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive cisplatin IV over 1 hour on day 1 and bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 76 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed pleural malignant mesothelioma, meeting 1 of the following criteria:

  * Recurrent disease after radical surgery
  * Disease not considered suitable for radical treatment
* Measurable or evaluable disease
* No clinical evidence of brain or leptomeningeal metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy > 12 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Creatinine clearance > 60 mL/min OR > 50 mL/min
* ALT and AST < 2.5 times upper limit of normal (ULN) (< 5 times ULN if liver metastases present)
* Bilirubin < 1.5 times ULN
* No concurrent secondary malignancy except carcinoma in situ of the cervix or adequately treated basal cell skin cancer
* No other malignancy treated within the past 5 years

  * Melanoma, breast cancer, or hypernephroma treated within the past 5 years and without recurrence are allowed
* No uncontrolled or severe cardiovascular disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class III-IV heart failure
  * Uncontrolled angina
  * Clinically significant pericardial disease or cardiac amyloidosis
* No infiltrative pulmonary or pericardial disease
* No preexisting peripheral neuropathy
* No known or suspected allergy or intolerance to boron, mannitol, or heparin, if an indwelling catheter is used
* No psychological, familial, sociological, or geographical condition that would preclude protocol compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy for mesothelioma
* No other concurrent antineoplastic agents except medications that may have antineoplastic activity but are taken for other reasons (e.g., megestrol acetate, cyclooxygenase-2 inhibitors, or bisphosphonates)
* No other concurrent experimental agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-02; Primary Completion 2010-04 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 18 weeks

SECONDARY OUTCOMES:
Overall objective response rate
Symptomatic response rate
Safety as measured by NCI CTCAE v3.0 and the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity questionnaire
Duration of PFS
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Mary O'Brien, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - Surrey, Sutton, England, United Kingdom

REFERENCES:
- [Derived] Walter RFH, Sydow SR, Berg E, Kollmeier J, Christoph DC, Christoph S, Eberhardt WEE, Mairinger T, Wohlschlaeger J, Schmid KW, Mairinger FD. Bortezomib sensitivity is tissue dependent and high expression of the 20S proteasome precludes good response in malignant pleural mesothelioma. Cancer Manag Res. 2019 Sep 24;11:8711-8720. doi: 10.2147/CMAR.S194337. eCollection 2019. PMID 31576173
- [Derived] O'Brien ME, Gaafar RM, Popat S, Grossi F, Price A, Talbot DC, Cufer T, Ottensmeier C, Danson S, Pallis A, Hasan B, Van Meerbeeck JP, Baas P. Phase II study of first-line bortezomib and cisplatin in malignant pleural mesothelioma and prospective validation of progression free survival rate as a primary end-point for mesothelioma clinical trials (European Organisation for Research and Treatment of Cancer 08052). Eur J Cancer. 2013 Sep;49(13):2815-22. doi: 10.1016/j.ejca.2013.05.008. Epub 2013 Jun 20. PMID 23791541